CLINICAL TRIAL: NCT03511456
Title: An Effect and Safety Investigation on Percutaneous Endoscopic Lumbar Discectomy Technique to Remove Extraforaminal Disc Herniation at L5/S1 Segment Through 5th Transverse Process-facet Joint-sacrum Space
Brief Title: An Effect and Safety Observation on PELD Technique for Extraforaminal Disc Herniation at L5/S1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2018-022
Record Dates: First submitted 2018-03-28; First posted 2018-04-27 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2019-07

CONDITIONS: Neuralgia, Sciatic
Keywords: leg pain; waist pain; life quality
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FLLDH-PELD: Extraforaminal LDH patients received PELD operation
  Interventions: Procedure: PELD operation

INTERVENTIONS:
Procedure: PELD operation — Under local anesthesia, the introduction of 20G needles could be performed with fluoroscopy. After the needle traveled through TFS space, extremely care was needed to avoid nerve root injury.
  Discography was recommended. The following steps were performed as usual: the needle was replaced by a guide wire; a 9 mm incision was made in the skin; a tapered cannulated dilator was inserted along the guide wire; and finally a working cannula was inserted.
  The remove of disc was performed carefully under endoscope. The first step was to locate the annulus fibrosis of L5/S1 disc, then by using nerve dissector and bipolar elliquence, soft tissue including fat tissue, muscle and fibers of ligaments were pushed cephalad until the blue stained herniated disc was visible and removed.

SUMMARY:
43% or so of far lateral lumbar disc herniation (FLLDH) occurred at L5/S1, however, the surgical treatment is still quite challenging. We conducted a modified PELD technique that enable us to remove the extraforaminal herniated disc at L5/S1, through the anatomical space surrounded by transverse process, facet joint and sacrum (TFS space). This study is to this technique's effect and safety in a one year follow-up.

DETAILED DESCRIPTION:
30 cases diagnosed as extraforaminal disc herniation at the segment of Lumbar 5 / sacrum 1 (L5/S1) will be recruited in this investigation. All the patients will receive PELD operation following the strict procedure that penetrating through the TFS space. The pain score (VAS), physical ability (ODI score) and life quality (SF-36） will be evaluated one day before surgery and 2 days, 1 month and 3 months after the surgery. Any side effects such as infection, nerve damage, main blood vessel injury will be recorded.

The operation procedure must follow the following steps:

1. The patient was positioned prone.
2. The skin entry point was determined using axial MRI or CT images
3. During operation, with anterior posterior view of fluoroscopy, the longitudinal midline of lumbar spine on the skin (Line C), the line right across L5/S1 space (Line A) was marked on the skin. With lateral view, the line right across L5/S1 space was also marked on skin (Line B). The line A and B should be crossed. The final entry point on skin was on the Line A and away from midline with the distance measured on axial MRI or CT images as described above.
4. Local infiltration with 1% Lidocaine was applied to skin and deep fascia on the penetration path. The introduction of long 20G needles could be performed with continuous or intermittent fluoroscopy. The needle traveled through TFS space. Generally, the position just above S1 superior endplate has enough safe space from the existing nerve root that might be pushed downward by the protruded discs, so it is usually the target for needle puncture.

   Discography was strongly recommended to confirm diagnosis and distinguish the protruded disc from the surrounding soft tissue.
5. The following steps were performed as usual: the needle was replaced by a guide wire; a 9 mm incision was made in the skin at the entry site; a tapered cannulated dilator was inserted along the guide wire; and finally a beveled round working cannula of 8.0 mm in outer diameter was inserted, with the beveled tip touching the endplate of S1 and leaning against superior articular process of S1. If the TFS space is not big enough for working cannula, manual bone drills with blunt tip could be used to enlarge it.

Soft tissue including fat tissue, muscle and fibers of ligaments were pushed cephalad until the blue stained herniated disc was visible. Then the disc was removed. An absorbable gelatin sponge was impacted via the working cannula for hemostasis. A sterile dressing was applied with a one-point suture.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered with extraforaminal lumbar disc herniation at L5/S1
* Patients received percutaneous endoscopic lumbar discectomy

Exclusion Criteria:

* The diagnosis is not comply with the FLLDH
* patients not choose PELD operation
* patients unwilling to accept regular followup

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, diagnosed as extraforaminal lumbar disc herniation at L5/S1, and received the operation of percutaneous endoscopic lumbar discectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03-05 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-03-05 (Estimated)

PRIMARY OUTCOMES:
Pain score | The change of leg/waist pain before (1 day before operation) and post operation (2 days, 1 month and 3 months after operation).
  Pain evaluated by Visual Analogue Scale system. Using a scale ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" and the "agonizing pain" according to the patient's mark, providing a range of scores from 0-10. A higher score means intensifier pain. The effects of operation is based on the different VAS scores evaluated by pre- or post- surgical patients who described their pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-1), mild pain(2-5), moderate pain (6-8 mm), and severe pain (9-10).

SECONDARY OUTCOMES:
Life quality | The change of life quality before (1 day before operation) and post operation (2 days, 1 month and 3 months after operation).
  SF-36(The Short Form (36) Health Survey), a 36-item, patient-reported survey of patient health will be used for life quality evaluation. it consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health). The lower the score the more disability. The higher the score the less disability. The scores are compared pre- and post-operation.

OTHER OUTCOMES:
Physical functional ability | The change of physical functional ability before (1 day before operation) and post operation (2 days, 1 month and 3 months after operation).
  The life quality specially associated with LDP is evaluated by the Oswestry Disability Index (ODI), an index derived from the Oswestry Low Back Pain Questionnaire.The self-completed questionnaire contains ten topics including intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Patients choose 6 statements describing different potential scenarios in each topic. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Dehong Yang, MD,PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided